CLINICAL TRIAL: NCT01151774
Title: Validation of Transesophageal Echocardiography With to Measure Renal Resistive Index and to Predict Acute Kidney Injury
Brief Title: Validation of Transesophageal Echocardiography (TEE) to Measure Renal Resistive Index and to Predict Renal Injury
Status: Withdrawn | Type: Observational
Why Stopped: study entered twice, please see protocol 0120110047
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Other Study IDs: 0120100024
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Decreased Vascular Flow to Kidneys

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study doctors are trying to determine if the TEE measurements from your stomach are helpful in measuring the blood flow to the kidneys.

DETAILED DESCRIPTION:
The significant morbidity and mortality associated with acute kidney injury in critical care patients and after cardiac surgery is well-known. Studies have demonstrated between 1 to 30% postoperative mortality, and even higher rates of up to 70% when patients develop kidney failure and require dialysis. Even small increases in creatinine between 0 to 0.5 mg/dl can result in a greater than two-fold rise in 30-day mortality. Despite efforts to improve outcome, there has been no proven effective pharmacological interventions to treat acute kidney failure. Most recommendations are aimed at prevention by identifying high-risk patients, avoiding nephrotoxic drugs and minimizing intraoperative hypotensive insults.

There are few studies that have assessed renal blood flow using transesophageal echocardiography (TEE). Yang et al. examined the left renal artery of 60 patients using TEE during cardiac surgery and evaluated the feasibility of using TEE as a method to measure renal blood flow intraoperatively. Although they were only able to include 60% of the subjects due to technical difficulties, they did demonstrate less than 10% variability between measurements and therefore good reproducibility using TEE.

Renal blood flow may not be the best method to predict sufficient renal perfusion. Renal autoregulation is not preserved under general anesthesia even with the maintenance of adequate mean arterial blood pressure and cardiac output. Renal blood flow is further worsened by hemodilution and hypothermia. In addition, due to its pulsatile nature, the diameters of the renal arteries vary during the cardiac cycle and are a source of calculation error when determining renal blood flow as a function of renal blood velocity and arterial diameter.

Renal resistive index (RI) is a measure of intrarenal hemodynamics that is calculated using the blood flow velocities of segmental or intrarenal vessels and correlates with renal blood flow and renovascular resistance. The renal artery is not used because the flow varies and is inconsistent between systole and diastole. RI becomes elevated in pathological conditions and is associated with increasing creatinine, renal injury and dysfunction. As blood flow and creatinine clearance decrease through the renal vasculature, the resistive index increases. Resistive index may be a better gauge of renal dysfunction rather than renal blood flow because it is easier to assess and less dependent on obtaining a Doppler beam view that is oriented perfectly parallel to the blood flow. Because RI is a ratio of the renal blood flow velocities [RI = (peak systolic velocity - peak end diastolic velocity)/peak systolic velocity], the margin of error created by non-parallel Doppler beams cancels out.

Traditionally, resistive index is obtained by transabdominal Doppler ultrasonography (USG) although there have been transesophageal studies that have used RI as a secondary endpoint when examining renal blood flow. There is currently no technique that routinely uses TEE to intraoperatively monitor resistive index as a determination of adequate renal blood perfusion and an indication of renal compromise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with use of TEE as part of anesthetic plan as clinically determined by anesthesiologist
* Subjects with no contraindications to use of TEE or transabdominal doppler ultrasonography

Exclusion Criteria:

* Patients on hemodialysis/peritoneal dialysis
* Patients with a contraindication to use of TEE i.e.esophageal stricture, esophageal diverticulum, esophageal/gastric tumor, recent esophageal/gastric surgery or radiation to the chest
* Patients with a contraindication to use of transabdominal doppler ultrasonography
* Patients who are pregnant
* patients with esophageal varices
* Patient with bleeding disorders

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subject sample will consist of patients undergoing cardiac, vascular and major abdominal surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Validation of resistive index using TEE | Prior to surgical incision and postop

SECONDARY OUTCOMES:
Correlate post operative creatinine, BUN and GFR levels with intraoperative resistance index | Daily levels postoperatively to day 5 or discharge
  The investigators hypothesize that there is a correlation between abnormal TEE resistive index measures, intraoperative events and post operative renal function studies.

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Jackson, MD, JD, Principal Investigator — UMDNJ-NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No